CLINICAL TRIAL: NCT00676780
Title: Green Tea Extract and Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: Polyphenon Pharma (Unknown)
Responsible Party: Principal Investigator, Jerry McLarty, Professor, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H04-176
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer
Keywords: EGCG; polyphenols; biomarkers; prostate specific antigen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — polyphenon E; epigallocatechin gallate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ECGC Extract (Experimental): Single arm for a phase II study
  Interventions: Drug: Polyphenon E (EGCG)

INTERVENTIONS:
Drug: Polyphenon E (EGCG) — 4 capsules daily with a meal for the duration of the study
  Other Names: Polyphenon E

SUMMARY:
The purpose of the study is to see if a green tea extract can beneficially alter several markers of cancer risk and progression.

DETAILED DESCRIPTION:
To evaluate the short-term effects of a daily dose of Polyphenon E administered during the interval between prostate biopsy and radical prostatectomy in men with recently diagnosed prostate cancer. Endpoints will be changes in serum and tissue biomarkers related to progression of cancer.

The effect of Polyphenon E on tumor cell c-Met expression and phosphorylation is the primary objective. Secondary objectives include the effects on the other tissue and serum biomarkers. Evaluation of the safety and tolerability of Polyphenon E in this subject population is another objective.

1.1 Determine the effects of Polyphenon E on tumor cell c-Met expression and phosphorylation levels in patients with prostate cancer 1.2 Determine the effects of Polyphenon E on PI-3K activation in patients with prostate cancer 1.3 Determine the effects of Polyphenon E on MAPK activation in patients with prostate cancer 1.4 Determine the effects of Polyphenon E on expression levels of other proteins involved in motility and invasion such as Rho GTPases and extracellular proteinases in patients with prostate cancer 1.5 Determine the effects of Polyphenon E on markers of angiogenesis in patients with prostate cancer 1.6 Determine the effects of Polyphenon E on serum Prostate Specific Antigen (PSA) in patients with prostate cancer 1.7 Determine the effects of Polyphenon E on other serum markers: C-reactive protein (CRP), Insulin-Like Growth factor I (IGF-I), Insulin-like Growth Factor Binding Protein 3 (IGFBP-3), Hepatocyte Growth Factor HGF 1.8 Evaluate the safety and tolerability of Polyphenon E in this subject population

ELIGIBILITY:
Inclusion Criteria:

* recent biopsy positive for prostate cancer
* scheduled for prostatectomy
* must be able to swallow capsules
* Palpable mass by digital rectal examination (DRE)
* Ability to give informed consent and willingness to adhere to study protocol
* Age ≥ 18 years and less than 75

Exclusion Criteria:

* abnormal liver function
* Prior hormonal or surgical therapy for prostate cancer
* Liver or kidney problems that would interfere with metabolism of study drug
* Any condition that would hamper informed consent or ability to comply with study protocol
* Participation in another research study in the last three months
* Known malignancy at any site other than prostate
* Recent consumption of green tea (5 or more cups per day, within one week prior to biopsy)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2004-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry W McLarty, Ph.D., Principal Investigator — LSUHSC Shreveport
Locations (1):
- LSU Health Sciences Center, Shreveport, Louisiana, United States

REFERENCES:
- [Result] McLarty J, Bigelow RL, Smith M, Elmajian D, Ankem M, Cardelli JA. Tea polyphenols decrease serum levels of prostate-specific antigen, hepatocyte growth factor, and vascular endothelial growth factor in prostate cancer patients and inhibit production of hepatocyte growth factor and vascular endothelial growth factor in vitro. Cancer Prev Res (Phila). 2009 Jul;2(7):673-82. doi: 10.1158/1940-6207.CAPR-08-0167. Epub 2009 Jun 19. PMID 19542190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the urology clinic at LSU Health, Shreveport during the period of May 1, 2004 and February 20, 2008.
Pre-assignment Details: Exclusion criterias were determined before enrollment process.
Groups:
- ECGC Extract, Prostate Cancer: Single arm for a phase II study of EGCG extract and prostate cancer. Subjects are asked to take 4 polyphenol E (200mg) capsules daily with a meal for the duration of the study. Biomarkers are measured at baseline and then again at presurgery, the end point for the study.
Period: Overall Study
Arm/Group | ECGC Extract, Prostate Cancer
Started | 33
Completed | 26
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | ECGC Extract, Prostate Cancer
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 58.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Prostate Specific Antigen (PSA) of Prostate Cancer
Description: Change in serum prostate specific antigen (PSA) from baseline to post Polyphenol E treatment.
Time Frame: Baseline and 6 weeks
Population: The number of participants for analysis was determined per protocol.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- ECGC Extract: Single arm for a phase II study of the effects of Epigallocatechin Gallate (ECGC) polyphenol extract from green tea on biomarkers in patients with prostate cancer.
Arm/Group | ECGC Extract
Number analyzed (Participants) | 26
ng/mL | 0.86 [0.0425 to 2.4675]
Statistical Analysis 1: Comparison: ECGC Extract; Test type: Superiority or Other; p = 0.027, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Serum Vascular Endothelial Growth Factor (VEGF) and Prostate Cancer.
Description: Change in serum vascular endothelial growth factor (VEGF) from baseline to post Polyphenol E treatment.
Time Frame: Baseline and 6 weeks.
Population: The number of participants for analysis was determined per protocol.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- ECGC Extract: Single arm for a phase II study of the effects of ECGC polyphenol extract from green tea on biomarkers in patients with prostate cancer.
Arm/Group | ECGC Extract
Number analyzed (Participants) | 26
pg/mL | 26.8 [-6.315 to 123.38]
Statistical Analysis 1: Comparison: ECGC Extract; Test type: Superiority or Other; p = 0.023, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in Serum Hepatocyte Growth Factor (HGF) and Prostate Cancer.
Description: Change in serum hepatocyte growth factor (HGF) from baseline to post Polyphenol E treatment.
Time Frame: Baseline and 6 weeks
Population: Number of participants for analysis was determined per protocol.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- ECGC Extract: Epigallocatechin Gallate (ECGC) Single arm for a phase II study.
Arm/Group | ECGC Extract
Number analyzed (Participants) | 26
pg/mL | 96.67 [27.0837 to 358.7475]
Statistical Analysis 1: Comparison: ECGC Extract; Null hypothesis is no change, i.e. median change = 0.0; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | ECGC Extract, Prostate Cancer
Serious Adverse Events (participants affected / at risk) | 1/33
Other Adverse Events (participants affected / at risk) | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECGC Extract, Prostate Cancer (N=33)
Myocardial Infarction (Cardiac disorders) | 1 (1) — Subject suffered a heart attack prior to surgery procedure. Determined to be not related to study drug.

LIMITATIONS AND CAVEATS:
Patient compliance was an issue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No